CLINICAL TRIAL: NCT00411073
Title: A Study to Evaluate the Effect of Repeat Oral Doses of Darapladib on Cardiac Conduction as Compared to Placebo and a Single Oral Dose of Moxifloxacin
Brief Title: Study Of The Effects Of SB 480848 (Darapladib) On The Electrical Conduction Of The Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SB 480848/035
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Atherosclerosis
Keywords: darapladib; moxifloxacin; QT study
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Darapladib

SUMMARY:
This is a study to assess the effects of darapladib on the cardiac conduction of the heart as compared to placebo and moxifloxacin. This a four period crossover design with each period lasting about 10 days. There will be a 7 to 10 day wash out in between each period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Body weight greater than 50 kg (110 lbs) and a body mass index between 19 and 30
* Signed and dated written informed consent prior to admission to the study
* Subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Exclusion Criteria:

* cardiac abnormalities
* history of asthma or severe allergic reactions
* history of alcohol or drug abuse
* use of prescription or non-prescription drugs or vitamins or herbal supplements
* history of cholecystectomy or biliary tract disease
* pregnant or nursing women
* history of allergy to the study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-12

PRIMARY OUTCOMES:
Change in QTc interval as compared to placebo and moxifloxacin | throughout the study

SECONDARY OUTCOMES:
Change in ECG parameters as compared to placebo and moxifloxacin | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: SB 480848/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SB 480848/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SB 480848/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SB 480848/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SB 480848/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SB 480848/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SB 480848/035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register